CLINICAL TRIAL: NCT07261865
Title: Identifying Diabetes and Impaired Glucose Tolerance in ICU Patients and Assessing Their Impact on Organ Failure and Outcome.
Brief Title: Identifying Diabetes and Impaired Glucose Tolerance in ICU Patients
Acronym: DISCOVER
Status: Recruiting | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Collaborators: Frisius Medisch Centrum (Other)
Responsible Party: Principal Investigator, Jill Moser, Assistant Professor, University Medical Center Groningen
Other Study IDs: 20548
Record Dates: First submitted 2025-09-29; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Diabetes (DM); Critical Illness
Keywords: Critical Illness; Diabetes; DISCOVER
MeSH Terms: conditions — Diabetes Mellitus; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In the Netherlands, patients admitted to the ICU are classified as having diabetes based on whether their medical records indicate glucose management medication use (Dutch National Intensive Care Evaluation (NICE) Registry). However, this approach does not identify patients with 1) undiagnosed diabetes, 2) uncontrolled diabetes, 3) patients managing their condition through lifestyle modifications, or 4) individuals with prediabetes, which is considered an early stage of diabetes. Consequently, this may lead to an underestimation of the "true" prevalence of chronic dysglycaemia among ICU patients and as a result the impact of various glycaemic states on acute outcomes remain underexplored.

DETAILED DESCRIPTION:
Diabetes is one of the most common comorbidities among patients admitted to the intensive care unit. Previous studies have found that patients with diabetes are at higher risk of severe complications including infections, delayed wound healing, cardiovascular events and ultimately death while in the ICU.

In the Netherlands, patients admitted to the ICU are classified as having diabetes based on whether their medical records indicate glucose management medication use (Dutch National Intensive Care Evaluation (NICE) Registry). However, this approach does not identify patients with 1) undiagnosed diabetes, 2) uncontrolled diabetes, 3) patients managing their condition through lifestyle modifications, or 4) individuals with prediabetes, which is considered an early stage of diabetes. Consequently, this may lead to an underestimation of the prevalence of chronic dysglycaemia among ICU patients. Therefore, the "true" prevalence and impact of various glycaemic states in ICU patients and how they influence acute and long-term outcomes remain underexplored. Within the general Dutch population, diabetes is diagnosed in 7% of individuals, while approximately 30% of those aged over 45 have prediabetes. In the ICU, 17% of admitted patients require medication for diabetes management, highlighting a higher prevalence compared to the general population's 7%. Given that most patients (~87%) admitted to the ICU are older than 45 years, it is likely that the prevalence of prediabetes is elevated in ICU patients as well. It is essential to avoid underestimating the incidence of diabetes and impaired glucose tolerance to ensure that patients are managed properly during ICU stay and importantly after leaving the ICU. Diabetes diagnosis typically relies on (fasting) glucose levels yet diagnosing diabetes in ICU patients poses challenges due to stress and acute illness impacting blood glucose levels, leading to stress-induced hyperglycaemia. The investigators found that upon admission to the ICU, 77% of patients without diabetes exhibited high blood glucose levels, with 20% of these patients experiencing severe hyperglycaemia. The underlying cause of this hyperglycaemia is currently uncertain, but it may stem from acute critical illness, the effect of medications, previously undiagnosed diabetes or prediabetes, or a combination of these factors.

Since the investigators are currently unable to accurately determine if patients entering the ICU have diabetes or prediabetes using standard glucose measurements, measuring glycated haemoglobin (HbA1c) which reflects the average blood glucose levels over the past two or three months may be an alternative method which together with anthropometric, glycaemic parameters, and other metabolic traits will assist in assessing the risk of associated complications and the impact on organ injury. Given the rising incidence of diabetes in the general population, there is an increasing likelihood that a greater number of individuals will be admitted to the ICU with diabetes and prediabetes in the coming years. Moreover, the prevalence and impact of various glycaemic states in ICU patients and how they influence acute critical illness outcomes remain underexplored.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients admitted to the ICU

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients admitted to the ICU
Sampling Method: Non-Probability Sample
Enrollment: 4395 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
What is the prevalence of the various dysglycemic states in patients admitted to the ICU? | Day 1
  HbA1c 6%=normal, 6-6.4%=prediabetes, >6.5%=diabetes
What is the impact of chronic hyperglycemic states on acute (ICU mortality and organ injury) and long-term outcomes? | Up to 1 year
  ICU mortality, organ injury during ICU stay (Acute Kidney Injury defined by the KDIGO criteria), and 1-year mortality

CONTACTS AND LOCATIONS:
Overall Officials: Jill Moser, PhD, Principal Investigator — University Medical Center Groningen
Locations (2):
- Netherlands (2):
  - Frisius MC, Leeuwarden, Provincie Friesland
  - University Medical Center Groningen, Groningen, Provincie Groningen

REFERENCES:
- [Background] Luethi N, Cioccari L, Tanaka A, Kar P, Giersch E, Deane AM, Martensson J, Bellomo R. Glycated Hemoglobin A1c Levels Are Not Affected by Critical Illness. Crit Care Med. 2016 Sep;44(9):1692-4. doi: 10.1097/CCM.0000000000001656. PMID 26977855
- [Background] Yong PH, Weinberg L, Torkamani N, Churilov L, Robbins RJ, Ma R, Bellomo R, Lam QT, Burns JD, Hart GK, Lew JF, Martensson J, Story D, Motley AN, Johnson D, Zajac JD, Ekinci EI. The Presence of Diabetes and Higher HbA1c Are Independently Associated With Adverse Outcomes After Surgery. Diabetes Care. 2018 Jun;41(6):1172-1179. doi: 10.2337/dc17-2304. Epub 2018 Mar 26. PMID 29581095
- [Background] Torkamani N, Churilov L, Robbins R, Jerums G, Beik V, Radcliffe N, Patterson S, Bellomo R, Burns J, Hart GK, Lam Q, Power DA, MacIsaac RJ, Johnson DF, Zajac J, Ekinci EI. Diabetes and higher HbA1c levels are independently associated with adverse renal outcomes in inpatients following multiple hospital admissions. J Diabetes Complications. 2020 Jan;34(1):107465. doi: 10.1016/j.jdiacomp.2019.107465. Epub 2019 Oct 22. PMID 31735639
- [Background] Michalia M, Kompoti M, Koutsikou A, Paridou A, Giannopoulou P, Trikka-Graphakos E, Clouva-Molyvdas P. Diabetes mellitus is an independent risk factor for ICU-acquired bloodstream infections. Intensive Care Med. 2009 Mar;35(3):448-54. doi: 10.1007/s00134-008-1288-0. Epub 2008 Sep 20. PMID 18807006
- [Background] Carpenter DL, Gregg SR, Xu K, Buchman TG, Coopersmith CM. Prevalence and Impact of Unknown Diabetes in the ICU. Crit Care Med. 2015 Dec;43(12):e541-50. doi: 10.1097/CCM.0000000000001353. PMID 26465219